CLINICAL TRIAL: NCT04630782
Title: Precision Medicine in Systemic Sclerosis Gastrointestinal Disease: Evaluating Imaging and Stool Biomarkers for Differentiating Disease Stages and Treatment Responses
Brief Title: Evaluating Gut Imaging and Stool Biomarkers in Patients With Scleroderma-associated Gastrointestinal Disease
Acronym: Pre Med SSc GI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); Tan Tock Seng Hospital (Other); Changi General Hospital (Other); Sengkang General Hospital (Other); National University of Singapore (Other); Nanyang Technological University (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: PM-SScGI-01
Record Dates: First submitted 2020-03-12; First posted 2020-11-16 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Systemic Sclerosis; Imaging, Diagnostic; MRI Scans; PET-MRI Scan
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool and urine samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: The investigators will compare PET-MRI imaging and stool biomarkers between patients with VEDOSS/early SSc (n=40) and those with late SSc (n=20) not on immunosuppressive treatment.
  Participants will undergo a PET-MRI scan once at baseline.
  Interventions: Diagnostic Test: PET-MRI scan
- Aim 2: In early SSc patients (n=35), the investigators will determine change in biomarker levels from pre-treatment baseline to 6 months (primary end-point) and 12-months (secondary end-point) following MMF treatment.
  Participants will undergo PET-MRI scans at baseline, 6-month and 12-month.
  Interventions: Diagnostic Test: PET-MRI scan
- Exploratory aim: In patients with VEDOSS/early SSc (n=15) not on immunosuppressive treatment, the investigators will characterize imaging and stool biomarker changes over one year.
  Participants will undergo PET-MRI scans at baseline and 12-month.
  Interventions: Diagnostic Test: PET-MRI scan

INTERVENTIONS:
Diagnostic Test: PET-MRI scan — Participants will be scanned centrally at Clinical Imaging Research Centre (CIRC, Singapore), on a Biograph mMR PET-MR scanner. Combined FDG-PET-MRI scan is critical for co-registration of peristaltic bowel for optimal image quality. The oesophagus to anorectum will be imaged. The PET-MRI scan starts 60 minutes post-FDG injection of 6mCi and immediately after injecting 10mg hyoscine butylbromide to reduce peristalsis. MRI sequences are non-contrast.

SUMMARY:
Systemic sclerosis (SSc) is characterized by autoimmunity and vasculopathy resulting in fibrosis of the skin and internal organs including the Gastrointestinal (GI) tract. Key unmet clinical needs are the availability of non-invasive biomarkers for early diagnosis of SSc-GI, further characterization of different stages of SSc-GI and SSc-GI treatment response. The investigators propose combining MRI FDG-PET with MRI T1-MOLLI mapping, which has been applied to cardiac imaging to quantify histologically correlated cardiac fibrosis. T1-MOLLI enables detection and quantification of diffuse fibrosis without the need for contrast.

Aim 1: FDG-PET-MRI imaging (primary biomarker) and stool markers (secondary biomarker) will be compared between patients with VEDOSS/early SSc and those with late SSc not on immunosuppressive treatment.

Aim 2: Evaluation of change in biomarker levels from pre-treatment baseline to 6 months (primary end-point) and 12-months (secondary end-point) following MMF treatment, in early SSc patients

Using precision medicine approach in diagnosis and treatment evaluation, the investigators anticipate that this study will contribute significantly to advance management strategies for, and improve outcomes of SSc-GI disease.

DETAILED DESCRIPTION:
1. Aim 1 Determine if FDG-PET-MRI imaging biomarkers differentiate patients with VEDOSS/ early SSc (predominantly inflammatory) from those with late SSc (predominantly fibrosis). Stool markers will be used as secondary biomarkers supporting inflammation.

   Study design: cross-sectional; The investigators will compare biomarkers between patients with VEDOSS/early SSc and those with late SSc not on immunosuppressive treatment.
2. Aim 2 Evaluate FDG-PET-MRI imaging biomarker change over a 6- and 12-month treatment period with mycophenolate mofetil (MMF) in patients with early SSc. Stool markers will be used as secondary biomarkers supporting inflammation.

   Study design: longitudinal; In early SSc patients, the investigators will determine change in biomarker levels from pre-treatment baseline to 6 months (primary end-point) and 12-months (secondary end-point) following MMF treatment.
3. Exploratory Aim: In patients with VEDOSS/early SSc not on immunosuppressive treatment, the investigators will characterize imaging and stool biomarker changes over one year.

ELIGIBILITY:
Inclusion Criteria:

(i) ≥ 21 years old (ii) SSc fulfilling the American College of Rheumatology/European League Against Rheumatism (EULAR) 2013 criteria or VEDOSS fulfilling proposed criteria by EULAR

Aim 1 subject stratification:

(i) VEDOSS/ early SSc (≤3 years) or late SSc (> 5 years), with disease duration defined from onset of first non-Raynaud's symptom (ii) Not on any immunosuppressive treatment or prednisolone >10 mg /day 8 weeks before recruitment

Aim 2 subject stratification:

(i) early SSc (≤3 years) and (ii) starting on immunosuppressive treatment either

1. MMF + Prednisolone or
2. Other immunosuppressive treatment in combination with MMF + Prednisolone

Exploratory aim subject stratification:

(i) VEDOSS or early SSc (≤3 years) with disease duration defined from onset of first non-Raynaud's symptom (ii) Not on any immunosuppressive treatment or prednisolone >10 mg /day 8 weeks before recruitment

Exclusion Criteria:

(i) Lactating or pregnancy (ii) Allergy or contraindications to hyoscine butylbromide (e.g. myasthenia gravis, prostatic enlargement with urinary retention, clinically significant GI obstruction or ileus) (iii) Contraindications to MRI (iv) Infections 4 weeks before baseline measurements (v) On antibiotics 4 weeks before baseline measurements, unless given for treatment of small intestinal bacterial overgrowth (SIBO), a complication of SSc.

(vi) Malignancy or suspected malignancy within the last 2 years (vii) Diabetes on treatment

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Singapore General Hospital, National University Hospital, Tan Tock Seng Hospital, Changi General Hospital and Sengkang General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory or fibrosis FDG-PET-MRI imaging biomarkers in VEDOSS/early SSc or late SSc patients not on immunosuppresive treatment | Baseline
  PET-MRI imaging biomarkers: Inflammatory biomarker: PET SUV tissue to background ratio (TBR); fibrosis biomarker: native T1-MOLLI value.
Inflammatory biomarkers on FDG-PET-MRI imaging after 6 months (primary endpoint) and 12 months (secondary endpoint) of Mycophenolate mofetil treatment. | Baseline, 6-month and 12-month
  Change in PET SUV TBR from baseline at 6 months (Primary endpoint) and 12 months (secondary endpoint) following Mycophenolate mofetil treatment

SECONDARY OUTCOMES:
FDG-PET-MRI imaging over one year in patients with VEDOSS/early SSc not on immunosuppresive treatment | Baseline and 12-month
  Change in PET SUV TBR, Native T1-MOLLI value, GIT score from baseline at 12 months.
Stool biomarkers | baseline, 6 and 12 months
  Faecal-calprotectin, stool microbiota diversity, relative abundance according to taxonomic classifications.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Low, Principal Investigator — Singapore General Hospital
Locations (5):
- Singapore (5):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steen VD, Medsger TA. Changes in causes of death in systemic sclerosis, 1972-2002. Ann Rheum Dis. 2007 Jul;66(7):940-4. doi: 10.1136/ard.2006.066068. Epub 2007 Feb 28. PMID 17329309
- [Background] Barnes J, Mayes MD. Epidemiology of systemic sclerosis: incidence, prevalence, survival, risk factors, malignancy, and environmental triggers. Curr Opin Rheumatol. 2012 Mar;24(2):165-70. doi: 10.1097/BOR.0b013e32834ff2e8. PMID 22269658
- [Background] Ng X, Thumboo J, Low AH. Validation of the scleroderma health assessment questionnaire and quality of life in English and Chinese-speaking patients with systemic sclerosis. Int J Rheum Dis. 2012 Jun;15(3):268-76. doi: 10.1111/j.1756-185X.2012.01731.x. Epub 2012 Apr 29. PMID 22709488
- [Background] Santosa A, Tan CS, Teng GG, Fong W, Lim A, Law WG, Chan G, Ng SC, Low A. Lung and gastrointestinal complications are leading causes of death in SCORE, a multi-ethnic Singapore systemic sclerosis cohort. Scand J Rheumatol. 2016 Nov;45(6):499-506. doi: 10.3109/03009742.2016.1153141. Epub 2016 May 27. PMID 27232525
- [Background] Marie I, Ducrotte P, Denis P, Menard JF, Levesque H. Small intestinal bacterial overgrowth in systemic sclerosis. Rheumatology (Oxford). 2009 Oct;48(10):1314-9. doi: 10.1093/rheumatology/kep226. Epub 2009 Aug 20. PMID 19696066
- [Background] Lepri G, Guiducci S, Bellando-Randone S, Giani I, Bruni C, Blagojevic J, Carnesecchi G, Radicati A, Pucciani F, Marco MC. Evidence for oesophageal and anorectal involvement in very early systemic sclerosis (VEDOSS): report from a single VEDOSS/EUSTAR centre. Ann Rheum Dis. 2015 Jan;74(1):124-8. doi: 10.1136/annrheumdis-2013-203889. Epub 2013 Oct 15. PMID 24130266
- [Background] Avouac J, Fransen J, Walker UA, Riccieri V, Smith V, Muller C, Miniati I, Tarner IH, Randone SB, Cutolo M, Allanore Y, Distler O, Valentini G, Czirjak L, Muller-Ladner U, Furst DE, Tyndall A, Matucci-Cerinic M; EUSTAR Group. Preliminary criteria for the very early diagnosis of systemic sclerosis: results of a Delphi Consensus Study from EULAR Scleroderma Trials and Research Group. Ann Rheum Dis. 2011 Mar;70(3):476-81. doi: 10.1136/ard.2010.136929. Epub 2010 Nov 15. PMID 21081523
- [Background] McFarlane IM, Bhamra MS, Kreps A, Iqbal S, Al-Ani F, Saladini-Aponte C, Grant C, Singh S, Awwal K, Koci K, Saperstein Y, Arroyo-Mercado FM, Laskar DB, Atluri P. Gastrointestinal Manifestations of Systemic Sclerosis. Rheumatology (Sunnyvale). 2018;8(1):235. doi: 10.4172/2161-1149.1000235. Epub 2018 Mar 30. PMID 30057856
- [Background] Bruni C, Frech T, Manetti M, Rossi FW, Furst DE, De Paulis A, Rivellese F, Guiducci S, Matucci-Cerinic M, Bellando-Randone S. Vascular Leaking, a Pivotal and Early Pathogenetic Event in Systemic Sclerosis: Should the Door Be Closed? Front Immunol. 2018 Sep 7;9:2045. doi: 10.3389/fimmu.2018.02045. eCollection 2018. PMID 30245695
- [Background] Kawaguchi Y, Nakamura Y, Matsumoto I, Nishimagi E, Satoh T, Kuwana M, Sumida T, Hara M. Muscarinic-3 acetylcholine receptor autoantibody in patients with systemic sclerosis: contribution to severe gastrointestinal tract dysmotility. Ann Rheum Dis. 2009 May;68(5):710-4. doi: 10.1136/ard.2008.096545. Epub 2008 Sep 1. PMID 18762475
- [Background] Singh J, Mehendiratta V, Del Galdo F, Jimenez SA, Cohen S, DiMarino AJ, Rattan S. Immunoglobulins from scleroderma patients inhibit the muscarinic receptor activation in internal anal sphincter smooth muscle cells. Am J Physiol Gastrointest Liver Physiol. 2009 Dec;297(6):G1206-13. doi: 10.1152/ajpgi.00286.2009. Epub 2009 Sep 24. PMID 19779020
- [Background] Manetti M, Neumann E, Muller A, Schmeiser T, Saar P, Milia AF, Endlicher E, Roeb E, Messerini L, Matucci-Cerinic M, Ibba-Manneschi L, Muller-Ladner U. Endothelial/lymphocyte activation leads to prominent CD4+ T cell infiltration in the gastric mucosa of patients with systemic sclerosis. Arthritis Rheum. 2008 Sep;58(9):2866-73. doi: 10.1002/art.23806. PMID 18759276
- [Background] Taroni JN, Martyanov V, Huang CC, Mahoney JM, Hirano I, Shetuni B, Yang GY, Brenner D, Jung B, Wood TA, Bhattacharyya S, Almagor O, Lee J, Sirajuddin A, Varga J, Chang RW, Whitfield ML, Hinchcliff M. Molecular characterization of systemic sclerosis esophageal pathology identifies inflammatory and proliferative signatures. Arthritis Res Ther. 2015 Jul 29;17:194. doi: 10.1186/s13075-015-0695-1. PMID 26220546
- [Background] Johnson ME, Pioli PA, Whitfield ML. Gene expression profiling offers insights into the role of innate immune signaling in SSc. Semin Immunopathol. 2015 Sep;37(5):501-9. doi: 10.1007/s00281-015-0512-6. Epub 2015 Jul 30. PMID 26223504
- [Background] Hinchcliff M, Huang CC, Wood TA, Matthew Mahoney J, Martyanov V, Bhattacharyya S, Tamaki Z, Lee J, Carns M, Podlusky S, Sirajuddin A, Shah SJ, Chang RW, Lafyatis R, Varga J, Whitfield ML. Molecular signatures in skin associated with clinical improvement during mycophenolate treatment in systemic sclerosis. J Invest Dermatol. 2013 Aug;133(8):1979-89. doi: 10.1038/jid.2013.130. Epub 2013 Mar 14. PMID 23677167
- [Background] Chakravarty EF, Martyanov V, Fiorentino D, Wood TA, Haddon DJ, Jarrell JA, Utz PJ, Genovese MC, Whitfield ML, Chung L. Gene expression changes reflect clinical response in a placebo-controlled randomized trial of abatacept in patients with diffuse cutaneous systemic sclerosis. Arthritis Res Ther. 2015 Jun 13;17(1):159. doi: 10.1186/s13075-015-0669-3. PMID 26071192
- [Background] Assassi S, Wang X, Chen G, Goldmuntz E, Keyes-Elstein L, Ying J, Wallace PK, Turner J, Zheng WJ, Pascual V, Varga J, Hinchcliff ME, Bellocchi C, McSweeney P, Furst DE, Nash RA, Crofford LJ, Welch B, Pinckney A, Mayes MD, Sullivan KM. Myeloablation followed by autologous stem cell transplantation normalises systemic sclerosis molecular signatures. Ann Rheum Dis. 2019 Oct;78(10):1371-1378. doi: 10.1136/annrheumdis-2019-215770. Epub 2019 Aug 7. PMID 31391177
- [Background] Taroni JN, Greene CS, Martyanov V, Wood TA, Christmann RB, Farber HW, Lafyatis RA, Denton CP, Hinchcliff ME, Pioli PA, Mahoney JM, Whitfield ML. A novel multi-network approach reveals tissue-specific cellular modulators of fibrosis in systemic sclerosis. Genome Med. 2017 Mar 23;9(1):27. doi: 10.1186/s13073-017-0417-1. PMID 28330499
- [Background] Papachristos DA, Nikpour M, Hair C, Stevens WM. Intravenous cyclophosphamide as a therapeutic option for severe refractory gastric antral vascular ectasia in systemic sclerosis. Intern Med J. 2015 Oct;45(10):1077-81. doi: 10.1111/imj.12883. PMID 26429218
- [Background] Raja J, Nihtyanova SI, Murray CD, Denton CP, Ong VH. Sustained benefit from intravenous immunoglobulin therapy for gastrointestinal involvement in systemic sclerosis. Rheumatology (Oxford). 2016 Jan;55(1):115-9. doi: 10.1093/rheumatology/kev318. Epub 2015 Aug 28. PMID 26320139
- [Background] Allanore Y, Distler O. Systemic sclerosis in 2014: Advances in cohort enrichment shape future of trial design. Nat Rev Rheumatol. 2015 Feb;11(2):72-4. doi: 10.1038/nrrheum.2014.222. Epub 2015 Jan 6. PMID 25561368
- [Background] Tashkin DP, Elashoff R, Clements PJ, Goldin J, Roth MD, Furst DE, Arriola E, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M; Scleroderma Lung Study Research Group. Cyclophosphamide versus placebo in scleroderma lung disease. N Engl J Med. 2006 Jun 22;354(25):2655-66. doi: 10.1056/NEJMoa055120. PMID 16790698
- [Background] Tashkin DP, Roth MD, Clements PJ, Furst DE, Khanna D, Kleerup EC, Goldin J, Arriola E, Volkmann ER, Kafaja S, Silver R, Steen V, Strange C, Wise R, Wigley F, Mayes M, Riley DJ, Hussain S, Assassi S, Hsu VM, Patel B, Phillips K, Martinez F, Golden J, Connolly MK, Varga J, Dematte J, Hinchcliff ME, Fischer A, Swigris J, Meehan R, Theodore A, Simms R, Volkov S, Schraufnagel DE, Scholand MB, Frech T, Molitor JA, Highland K, Read CA, Fritzler MJ, Kim GHJ, Tseng CH, Elashoff RM; Sclerodema Lung Study II Investigators. Mycophenolate mofetil versus oral cyclophosphamide in scleroderma-related interstitial lung disease (SLS II): a randomised controlled, double-blind, parallel group trial. Lancet Respir Med. 2016 Sep;4(9):708-719. doi: 10.1016/S2213-2600(16)30152-7. Epub 2016 Jul 25. PMID 27469583
- [Background] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083
- [Background] Furst DE, Braun-Moscovic Y, Khanna D. Points to consider for clinical trials of the gastrointestinal tract in systemic sclerosis. Rheumatology (Oxford). 2017 Sep 1;56(suppl_5):v4-v11. doi: 10.1093/rheumatology/kex195. PMID 28992166
- [Background] Soussan M, Nicolas P, Schramm C, Katsahian S, Pop G, Fain O, Mekinian A. Management of large-vessel vasculitis with FDG-PET: a systematic literature review and meta-analysis. Medicine (Baltimore). 2015 Apr;94(14):e622. doi: 10.1097/MD.0000000000000622. PMID 25860208
- [Background] Lenze F, Wessling J, Bremer J, Ullerich H, Spieker T, Weckesser M, Gonschorrek S, Kannengiesser K, Rijcken E, Heidemann J, Luegering A, Schober O, Domschke W, Kucharzik T, Maaser C. Detection and differentiation of inflammatory versus fibromatous Crohn's disease strictures: prospective comparison of 18F-FDG-PET/CT, MR-enteroclysis, and transabdominal ultrasound versus endoscopic/histologic evaluation. Inflamm Bowel Dis. 2012 Dec;18(12):2252-60. doi: 10.1002/ibd.22930. Epub 2012 Feb 22. PMID 22359277
- [Background] Versari A, Pipitone N, Casali M, Jamar F, Pazzola G. Use of imaging techniques in large vessel vasculitis and related conditions. Q J Nucl Med Mol Imaging. 2018 Mar;62(1):34-39. doi: 10.23736/S1824-4785.17.03044-8. Epub 2017 Nov 22. PMID 29166756
- [Background] Einspieler I, Thurmel K, Pyka T, Eiber M, Wolfram S, Moog P, Reeps C, Essler M. Imaging large vessel vasculitis with fully integrated PET/MRI: a pilot study. Eur J Nucl Med Mol Imaging. 2015 Jun;42(7):1012-24. doi: 10.1007/s00259-015-3007-8. Epub 2015 Apr 16. PMID 25876704
- [Background] Beiderwellen K, Kinner S, Gomez B, Lenga L, Bellendorf A, Heusch P, Umutlu L, Langhorst J, Ruenzi M, Gerken G, Bockisch A, Lauenstein TC. Hybrid imaging of the bowel using PET/MR enterography: Feasibility and first results. Eur J Radiol. 2016 Feb;85(2):414-21. doi: 10.1016/j.ejrad.2015.12.008. Epub 2015 Dec 17. PMID 26781147
- [Background] Pellino G, Nicolai E, Catalano OA, Campione S, D'Armiento FP, Salvatore M, Cuocolo A, Selvaggi F. PET/MR Versus PET/CT Imaging: Impact on the Clinical Management of Small-Bowel Crohn's Disease. J Crohns Colitis. 2016 Mar;10(3):277-85. doi: 10.1093/ecco-jcc/jjv207. Epub 2015 Nov 15. PMID 26574490
- [Background] Catalano OA, Gee MS, Nicolai E, Selvaggi F, Pellino G, Cuocolo A, Luongo A, Catalano M, Rosen BR, Gervais D, Vangel MG, Soricelli A, Salvatore M. Evaluation of Quantitative PET/MR Enterography Biomarkers for Discrimination of Inflammatory Strictures from Fibrotic Strictures in Crohn Disease. Radiology. 2016 Mar;278(3):792-800. doi: 10.1148/radiol.2015150566. Epub 2015 Oct 5. PMID 26436860
- [Background] Marchesseau S, Ng SA, Wang YT, Xie W, Ng DC, Totman JJ, Low AHL. 18F-FDG PET-MRI with T1 MOLLI mapping to detect systemic sclerosis bowel inflammation and fibrosis. Eur J Radiol. 2018 Aug;105:289-295. doi: 10.1016/j.ejrad.2018.06.022. Epub 2018 Jun 26. PMID 30017295
- [Background] Freiman M, Perez-Rossello JM, Callahan MJ, Bittman M, Mulkern RV, Bousvaros A, Warfield SK. Characterization of fast and slow diffusion from diffusion-weighted MRI of pediatric Crohn's disease. J Magn Reson Imaging. 2013 Jan;37(1):156-63. doi: 10.1002/jmri.23781. Epub 2012 Aug 24. PMID 22927342
- [Background] Zhang MC, Li XH, Huang SY, Mao R, Fang ZN, Cao QH, Zhang ZW, Yan X, Chen MH, Li ZP, Sun CH, Feng ST. IVIM with fractional perfusion as a novel biomarker for detecting and grading intestinal fibrosis in Crohn's disease. Eur Radiol. 2019 Jun;29(6):3069-3078. doi: 10.1007/s00330-018-5848-6. Epub 2018 Dec 13. PMID 30547200
- [Background] Le Bihan D. What can we see with IVIM MRI? Neuroimage. 2019 Feb 15;187:56-67. doi: 10.1016/j.neuroimage.2017.12.062. Epub 2017 Dec 22. PMID 29277647
- [Background] Volkmann ER. Intestinal microbiome in scleroderma: recent progress. Curr Opin Rheumatol. 2017 Nov;29(6):553-560. doi: 10.1097/BOR.0000000000000429. PMID 28719392
- [Background] Volkmann ER, Hoffmann-Vold AM, Chang YL, Jacobs JP, Tillisch K, Mayer EA, Clements PJ, Hov JR, Kummen M, Midtvedt O, Lagishetty V, Chang L, Labus JS, Molberg O, Braun J. Systemic sclerosis is associated with specific alterations in gastrointestinal microbiota in two independent cohorts. BMJ Open Gastroenterol. 2017 Apr 1;4(1):e000134. doi: 10.1136/bmjgast-2017-000134. eCollection 2017. PMID 28761687
- [Background] Ishikawa D, Sasaki T, Osada T, Kuwahara-Arai K, Haga K, Shibuya T, Hiramatsu K, Watanabe S. Changes in Intestinal Microbiota Following Combination Therapy with Fecal Microbial Transplantation and Antibiotics for Ulcerative Colitis. Inflamm Bowel Dis. 2017 Jan;23(1):116-125. doi: 10.1097/MIB.0000000000000975. PMID 27893543
- [Background] Low AHL, Teng GG, Pettersson S, de Sessions PF, Ho EXP, Fan Q, Chu CW, Law AHN, Santosa A, Lim AYN, Wang YT, Haaland B, Thumboo J. A double-blind randomized placebo-controlled trial of probiotics in systemic sclerosis associated gastrointestinal disease. Semin Arthritis Rheum. 2019 Dec;49(3):411-419. doi: 10.1016/j.semarthrit.2019.05.006. Epub 2019 May 23. PMID 31208714
- [Background] Bjerrum JT, Wang Y, Hao F, Coskun M, Ludwig C, Gunther U, Nielsen OH. Metabonomics of human fecal extracts characterize ulcerative colitis, Crohn's disease and healthy individuals. Metabolomics. 2015;11:122-133. doi: 10.1007/s11306-014-0677-3. Epub 2014 Jun 1. PMID 25598765
- [Background] Waclawikova B, El Aidy S. Role of Microbiota and Tryptophan Metabolites in the Remote Effect of Intestinal Inflammation on Brain and Depression. Pharmaceuticals (Basel). 2018 Jun 25;11(3):63. doi: 10.3390/ph11030063. PMID 29941795
- [Background] Andreasson K, Alrawi Z, Persson A, Jonsson G, Marsal J. Intestinal dysbiosis is common in systemic sclerosis and associated with gastrointestinal and extraintestinal features of disease. Arthritis Res Ther. 2016 Nov 29;18(1):278. doi: 10.1186/s13075-016-1182-z. PMID 27894337
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] Khanna D, Furst DE, Clements PJ, Allanore Y, Baron M, Czirjak L, Distler O, Foeldvari I, Kuwana M, Matucci-Cerinic M, Mayes M, Medsger T Jr, Merkel PA, Pope JE, Seibold JR, Steen V, Stevens W, Denton CP. Standardization of the modified Rodnan skin score for use in clinical trials of systemic sclerosis. J Scleroderma Relat Disord. 2017 Jan-Apr;2(1):11-18. doi: 10.5301/jsrd.5000231. PMID 28516167
- [Background] Sprooten RTM, Lenaerts K, Braeken DCW, Grimbergen I, Rutten EP, Wouters EFM, Rohde GGU. Increased Small Intestinal Permeability during Severe Acute Exacerbations of COPD. Respiration. 2018;95(5):334-342. doi: 10.1159/000485935. Epub 2018 Jan 25. PMID 29393240
- [Background] Rizzetto L, Fava F, Tuohy KM, Selmi C. Connecting the immune system, systemic chronic inflammation and the gut microbiome: The role of sex. J Autoimmun. 2018 Aug;92:12-34. doi: 10.1016/j.jaut.2018.05.008. Epub 2018 Jun 1. PMID 29861127
- [Background] Khanna D, Hays RD, Maranian P, Seibold JR, Impens A, Mayes MD, Clements PJ, Getzug T, Fathi N, Bechtel A, Furst DE. Reliability and validity of the University of California, Los Angeles Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument. Arthritis Rheum. 2009 Sep 15;61(9):1257-63. doi: 10.1002/art.24730. PMID 19714600
- [Background] Low AHL, Xin X, Law WG, Teng GG, Santosa A, Lim A, Chan G, Ng SC, Thumboo J. Validation of the UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument 2.0 in English- and Chinese-speaking patients in a multi-ethnic Singapore systemic sclerosis cohort. Clin Rheumatol. 2017 Jul;36(7):1643-1648. doi: 10.1007/s10067-016-3529-x. Epub 2017 Jan 5. PMID 28058539
- [Background] Khanna D, Furst DE, Maranian P, Seibold JR, Impens A, Mayes MD, Clements PJ, Getzug T, Hays RD. Minimally important differences of the UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument. J Rheumatol. 2011 Sep;38(9):1920-4. doi: 10.3899/jrheum.110225. Epub 2011 Jul 1. PMID 21724699
- [Background] Korecka A, Dona A, Lahiri S, Tett AJ, Al-Asmakh M, Braniste V, D'Arienzo R, Abbaspour A, Reichardt N, Fujii-Kuriyama Y, Rafter J, Narbad A, Holmes E, Nicholson J, Arulampalam V, Pettersson S. Bidirectional communication between the Aryl hydrocarbon Receptor (AhR) and the microbiome tunes host metabolism. NPJ Biofilms Microbiomes. 2016 Aug 24;2:16014. doi: 10.1038/npjbiofilms.2016.14. eCollection 2016. PMID 28721249
- [Background] Thion MS, Low D, Silvin A, Chen J, Grisel P, Schulte-Schrepping J, Blecher R, Ulas T, Squarzoni P, Hoeffel G, Coulpier F, Siopi E, David FS, Scholz C, Shihui F, Lum J, Amoyo AA, Larbi A, Poidinger M, Buttgereit A, Lledo PM, Greter M, Chan JKY, Amit I, Beyer M, Schultze JL, Schlitzer A, Pettersson S, Ginhoux F, Garel S. Microbiome Influences Prenatal and Adult Microglia in a Sex-Specific Manner. Cell. 2018 Jan 25;172(3):500-516.e16. doi: 10.1016/j.cell.2017.11.042. Epub 2017 Dec 21. PMID 29275859
- [Background] Bjerrum JT, Steenholdt C, Ainsworth M, Nielsen OH, Reed MA, Atkins K, Gunther UL, Hao F, Wang Y. Metabonomics uncovers a reversible proatherogenic lipid profile during infliximab therapy of inflammatory bowel disease. BMC Med. 2017 Oct 16;15(1):184. doi: 10.1186/s12916-017-0949-7. PMID 29032767
- [Background] Rutten EPA, Lenaerts K, Buurman WA, Wouters EFM. Disturbed intestinal integrity in patients with COPD: effects of activities of daily living. Chest. 2014 Feb;145(2):245-252. doi: 10.1378/chest.13-0584. PMID 23928850
- [Background] Morrisroe K, Sudararajan V, Stevens W, Sahhar J, Zochling J, Roddy J, Proudman S, Nikpour M. Work productivity in systemic sclerosis, its economic burden and association with health-related quality of life. Rheumatology (Oxford). 2018 Jan 1;57(1):73-83. doi: 10.1093/rheumatology/kex362. PMID 29155994
- [Background] Forbes A, Marie I. Gastrointestinal complications: the most frequent internal complications of systemic sclerosis. Rheumatology (Oxford). 2009 Jun;48 Suppl 3:iii36-9. doi: 10.1093/rheumatology/ken485. PMID 19487222